CLINICAL TRIAL: NCT01246895
Title: Follow-up Study Evaluating The Long-Term Safety and Efficacy of BST-CarGel® and Microfracture In Repair of Focal Articular Cartilage Lesions on The Femoral Condyle (Extension Study of Protocols CG-CIP01-P & CG-CIP02-P)
Brief Title: Follow-Up Study Evaluating The Long Term Safety and Efficacy of BST-CarGel and Microfracture Repair of the Knee
Status: Completed | Type: Observational
Sponsor: Piramal Healthcare Canada Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CG-CIP04-P
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2016-11

CONDITIONS: Knee Injuries
Keywords: Cartilage repair; Cartilage; Knee; Knee Pain; Microfracture; Arthroscopy; Bone Marrow Stimulation; Chondrogenesis; Scaffold; Chitosan; Articular Cartilage Repair
MeSH Terms: conditions — Knee Injuries; Fractures, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Microfracture with BST-CarGel
  Interventions: Device: Microfracture with BST-CarGel
- Control: Microfracture without BST-CarGel
  Interventions: Device: Microfracture without BST-CarGel

INTERVENTIONS:
Device: Microfracture with BST-CarGel
  Groups: Experimental
Device: Microfracture without BST-CarGel
  Groups: Control

SUMMARY:
This follow-up study will evaluate the effects of BST-CarGel® application to a microfractured lesion (investigational) and microfracture alone (control) for up to 5 years from treatment in subjects, treated under Protocols CG-CIP01-P and CG-CIP02-P, and will serve as a post approval study for these Protocols, in support of a commercial application. The lesions treated under Protocols CG-CIP01-P and CG-CIP02-P were focal lesions of articular cartilage, grade 3 or 4 (either ICRS or Outerbridge classification) on the medial and lateral femoral condyles of the knee, and were classified as either acute or chronic.

DETAILED DESCRIPTION:
Cartilage repair currently remains a problematic orthopedic concern with no effective solution. The development of new surgical techniques or therapies is critical in meeting this medical need.

Clinical data regarding the long-term durability of repair tissue resulting from cartilage repair techniques such as microfracture, autologous chondrocyte implantation or mosaicplasty is lacking. Only two studies, one comparative and one uncontrolled, have examined long-term repair outcomes (over 4 years). These studies reinforced the concept that further studies are needed to identify a technique or product that will lead to long-term clinical benefit through improved cartilage repair efficacy.

BST-CarGel® is a medical device derived from chitosan applied to a microfractured lesion and has been shown to promote the quantity and quality of cartilage repair tissue in animals. The efficacy and safety of BST-CarGel® is currently being evaluated in humans as compared to the standard of care treatment, microfracture, in a 12 month international study in Canada, Europe and Korea under Protocols CG-CIP01-P and CG-CIP02-P. When these protocols were designed and carried out, the BST-CarGel® technology belonged to BioSyntech Canada Inc. Afterwards, the technology was acquired by Piramal Healthcare (Canada) Ltd. which is now the owner of the technology and the sponsor for this Extension Study CG-C1P04.

This follow-up study will evaluate the long-term effects (5 yrs) of BST-CarGel® + microfracture and microfracture alone in subjects treated in the pivotal and sub-studies.

All eligible subjects (maximum 80) who were treated under Protocols CG-CIP01-P and CG-CIP02-P and completed the required 12 month follow-up period will be asked to participate in this follow-up study.

The stratification from Protocols CG-CIP01-P and CG-CIP02-P (investigational site and lesion type) will be retained for the purposes of the follow-up study, and all third parties such as the MRI central reading facility will remain blinded to the treatment received under Protocols CG-CIP01-P and CG-CIP02-P.

Comparisons between the two treatment groups will be performed.

The following assessments will be done annually at years 3 and/or 4 and 5 post -treatment under Protocols CG-CIP01-P and CG-CIP02-P in subjects treated with BST-CarGel + microfracture or microfracture alone:

1. Analyses of tissue repair will be carried out based on the degree of lesion filling and quality of repair tissue using MRI
2. The general health status of subjects will be captured in the case report form (CRF) and will include the subject's overall health status, treated knee status, adverse events (AEs) and concomitant medications.
3. The assessment of the subject's knee pain, stiffness, functional ability and quality of life through self-assessment questionnaires (Western Ontario and McMaster Universities osteoarthritis index (WOMAC) and short-form-36 (SF-36v2)

ELIGIBILITY:
Inclusion Criteria:

* The subject was treated under Protocol CG-CIP01 or CG-CIP02 and completed 12 month follow-up period
* The subject has understood and signed a Research Ethics Board(REB) approved Informed Consent Form (ICF)

Exclusion Criteria:

* The subject was not treated under Protocol CG-CIP01-P or CG-CIP02-P
* The subject did not complete 12 month follow-up period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients that have been treated under either protocol CG-CIP01 or CG-CIP02
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Stanish, M.D, Principal Investigator — Orthopaedic and Sport Medicine - Dalhousie University
Locations (16):
- Canada (11):
  - University of Calgary Sports Medicine Centre, Calgary, Alberta
  - Simon Fraser Orthopaedic Fund, Royal Columbian Hospital, New Westminster, British Columbia
  - Joint Preservation Centre of British Columbia, Vancouver, British Columbia
  - Pan Am Clinic, Winnipeg, Manitoba
  - Orthopaedic and Sport Medicine Clinic of Nova Scotia, Halifax, Nova Scotia
  - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Sports Medicine Center, Carleton University, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Orthopaedics Research Office, Toronto, Ontario
  - Hospital Sacré-Coeur de Montréal, Montreal, Quebec
  - CHA-Pavillon Enfant-Jésus, Québec, Quebec
  - Hôpital Charles LeMoyne, Unité d'investigation non invasive, Québec, Quebec
- Spain (5):
  - FREMAP Centro de Prevención y Rehabilitatión, Majadahonda, Madrid
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Cirugia Ortopedica y Traumatologia, Medicina del Deporte, Gijón
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Result] Shive MS, Stanish WD, McCormack R, Forriol F, Mohtadi N, Pelet S, Desnoyers J, Methot S, Vehik K, Restrepo A. BST-CarGel(R) Treatment Maintains Cartilage Repair Superiority over Microfracture at 5 Years in a Multicenter Randomized Controlled Trial. Cartilage. 2015 Apr;6(2):62-72. doi: 10.1177/1947603514562064. PMID 26069709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible subjects who were treated under Protocol CG-CIP01-P and completed the required 12-month follow-up period were asked to participate in this follow-up study. Ultimately, 67 subjects signed an ICF to enter the study and the screening process.
Groups:
- Microfracture + BST-CarGel: Microfracture with BST-CarGel
- Microfracture Alone: Microfracture without BST-CarGel
Period: Overall Study
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
Started | 37 | 30
Completed | 34 | 26
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: Sample size determination for the 1-year trial was previously reported. All treated participants who enrolled in the extension study were included in the efficacy analyses, which were performed according to a preapproved statistical analysis plan.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (9.7) | 40.1 (10.1) | 36.8 (10.2)
Sex/Gender, Customized [Number; unit: participants]
  Male | 22 | 14 | 36
  Female | 12 | 12 | 24
  Withdrew/Withdrawn | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 26 | 56
  Spain | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Degree of Lesion Filling (%Fill) by Repair Tissue at Degree of Lesion Filling (%Fill) by Repair Tissue at 5 Years Through MRI.
Description: Degree of lesion filling (repair tissue volume) as measured by quantitative MRI at 5 Years post-treatment compared to the debrided lesion 1-month post-treatment (baseline).
Time Frame: 5 years
Population: 33 out of 34 BST-CarGel with percentage lesion filled measurement. 1 aberrant imaging datapoint from 1 patient out of 34 patients was removed from the Experimental group
Measure: Least Squares Mean (Standard Deviation); unit: Percentage of lesion filled (%)
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
Number analyzed (Participants) | 33 | 26
Percentage of lesion filled (%) | 93.79 (1.16) | 86.96 (2.85)
Statistical Analysis 1: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; Test type: Superiority or Other; p = 0.017, general estimating equations (GEE) — P-values were obtained using general estimating equations (GEE) for longitudinal analysis of repeated correlated measures; P-values were obtained using general estimating equations (GEE) for longitudinal analysis of repeated correlated measures

2. Primary Outcome: Repair Tissue Quality (T2 MRI)
Description: Tissue quality of the repair tissue as measured by T2 MRI as an index for collagen-based structure.
Time Frame: 5 years
Population: 5 aberrant imaging datapoint from 5 patients out of 34 patients were removed from the Experimental group and 4 aberrant imaging datapoint from 4 patients out of 34 patients were removed from the Control group
Measure: Least Squares Mean (Standard Deviation); unit: T2 relaxation time (ms)
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
Number analyzed (Participants) | 29 | 22
T2 relaxation time (ms) | 75.68 (5.25) | 90.41 (6.56)
Statistical Analysis 1: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; Test type: Superiority or Other; p = 0.026, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage Change From Baseline for Knee-related Pain, Stiffness and Function at 5 Years (WOMAC Parts A, B, C)
Description: The three sub-scales: 1) Pain, 2.) stiffness and 3.) function scores ranged from 0-10. Pain had 5 items and stiffness had 2 items, and function had 17 items. The total score for pain ranged from 0 no pain to 50 worst pain. The total score for stiffness ranged from 0 no stiffness to 20 worst stiffness. The total score for function raged from 0 no function to 170 worst function. A higher score indicates a better health state improvement.
Time Frame: 5 years
Population: 1 datapoint not made available from 1 patient out of 34 patients in the Experimental group
Measure: Least Squares Mean (Standard Deviation); unit: Percentage change
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
Number analyzed (Participants) | 33 | 26
Percentage change
  Pain at 5 year | -15.37 (1.47) | -16.56 (1.19)
  Stiffness at 5 year | -5.63 (0.72) | -6.68 (0.58)
  Physical Function at 5 year | -56.52 (4.57) | -62.10 (3.43)
Statistical Analysis 1: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; WOMAC subscale - Pain; Test type: Superiority or Other; p = 0.474, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; WOMAC subscale - Stiffness; Test type: Superiority or Other; p = 0.236, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; WOMAC subscale - Physical function; Test type: Superiority or Other; p = 0.326, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: The Number of Participants With Adverse Events Until 5 Years
Description: Safety was assessed by recording the number of participants with Adverse Events (AEs) and their severity from the time of ICF signing up to 5 years post-treatment.
Time Frame: 5 years
Population: Participants who experienced adverse events
Measure: Number; unit: participants
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
Number analyzed (Participants) | 34 | 26
participants
  Participants with AE's | 13 | 18
  Participants with unanticipated procedure-related | 1 | 0
  Participants with anticipated procedure-related AE | 1 | 2
  Participants with unanticipated device-related AEs | 1 | 0
  Participants with anticipated device-related AEs | 0 | 0
  Participants with serious adverse events SAEs | 1 | 0
  Participants discontinued from study because of an | 0 | 0
  Participant death over the 5-year follow up period | 0 | 0
Statistical Analysis 1: Comparison: Microfracture + BST-CarGel vs Microfracture Alone; Test type: Superiority or Other; p = 0.01, Physical count

5. Other Pre Specified Outcome: Percentage Change in Quality of Life Assessed Using the SF-36 Questionnaire.
Description: SF-36 v2 includes 2 aggregate measures-Physical and Mental components-derived from 8 subscales. Least squares means are adjusted for baseline. Higher positive scores indicate better results. Scoring ranges from 0 to 100%.
Time Frame: 1 and 5 years
Measure: Least Squares Mean (Standard Deviation); unit: Percent change from baseline
Groups:
- Expiremental: Microfracture with BST-CarGel
Arm/Group | Expiremental | Control
Number analyzed (Participants) | 34 | 27
Percent change from baseline
  Physical component - Year 1 | 13.01 (1.43) | 14.37 (1.35)
  Physical component - Year 5 | 13.12 (1.63) | 14.48 (1.42)
  Mental component - Year 1 | 3.38 (1.42) | 0.49 (1.42)
  Mental component - Year 5 | 2.72 (1.30) | -0.17 (1.76)
Statistical Analysis 1: Comparison: Expiremental vs Control; SF-36 v2 Physical component; Test type: Superiority or Other; p = 0.478, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Expiremental vs Control; SF-36 v2 Mental component; Test type: Superiority or Other; p = 0.125, general estimating equations (GEE) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events collected from signature of ICF (follow-up study) to 5 year follow-up.
Description: The incidence of AEs, SAEs, and incidents have been summarized by SOC and preferred terms according to MedDRA preferred terminology for each treatment group, frequency, maximum severity, and relationship to procedure or device.
Arm/Group | Microfracture + BST-CarGel | Microfracture Alone
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/30
Other Adverse Events (participants affected / at risk) | 2/37 | 3/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microfracture + BST-CarGel (N=37) | Microfracture Alone (N=30)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microfracture + BST-CarGel (N=37) | Microfracture Alone (N=30)
LEFT KNEE THROBBING PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unanticipated procedure/device-related. Preferred Term: Arthralgia
LEFT KNEE MEDIAL CLICKING THAT INITIATES THROBBING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unanticipated procedure/device-related. Preferred Term: Arthralgia
PAIN LEFT KNEE/ ABOVE KNEE CAP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Anticipated procedure-related. Preferred Term: Arthralgia.
FEELING OF RIGHT KNEE GIVING OUT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Anticipated procedure-related. Preferred Term: Arthralgia.
RIGHT KNEE PAIN AFTER EXERCISE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Anticipated procedure-related. Preferred Term: Arthralgia
MIGRAINES (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Since the sample size was not predetermined, the statistical methods were used in a conditional fashion such that those that were determined to be invalid or inappropriate upon data review were discarded or replaced by more appropriate analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less